CLINICAL TRIAL: NCT03375567
Title: Global Response Assessment by Advanced Imaging and Myeloma Lesion Biopsies During Induction Therapy of Multiple Myeloma With Carfilzomib Lenalidomide Dexamethasone (CRD)
Brief Title: Global Response Assessment by Advanced Imaging and Myeloma Lesion Biopsies During Induction Therapy of Multiple Myeloma With Carfilzomib Lenalidomide Dexamethasone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000021421
Record Dates: First submitted 2017-12-12; First posted 2017-12-18 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: After patients are treated with Carfilzomib Lenalidomide Dexamethasone (CRD), lesion biopsies will be performed per usual care. Patients will have biopsies performed on lesions using a novel image guided technique.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Lesion Biopsies (Experimental): After patients are treated with Carfilzomib Lenalidomide Dexamethasone (CRD), lesion biopsies will be performed per usual care. Patients will have biopsies performed on lesions using a novel image guided technique.
  Interventions: Procedure: Guided Lesion Biopsies
- Standard Lesion Biopsies (Active Comparator): After patients are treated with Carfilzomib Lenalidomide Dexamethasone (CRD), lesion biopsies will be performed per usual care. Patients will have biopsies performed on lesions using a novel image guided technique.
  Interventions: Procedure: Standard Lesion Biopsies

INTERVENTIONS:
Procedure: Guided Lesion Biopsies — After patients are treated with Carfilzomib Lenalidomide Dexamethasone (CRD), lesion biopsies will be performed per usual care. Patients will have biopsies performed on lesions using a novel image guided technique.
  Arms: Guided Lesion Biopsies
Procedure: Standard Lesion Biopsies — After patients are treated with Carfilzomib Lenalidomide Dexamethasone (CRD), lesion biopsies will be performed per usual care. Patients will have biopsies performed on lesions using a novel image guided technique.
  Arms: Standard Lesion Biopsies

SUMMARY:
The primary objective of this study is to compare the detection rate of residual/refractory disease based on standard bone marrow biopsy versus guided myeloma lesion biopsy after induction therapy with carfilzomib, lenalidomide and dexamethasone regimen.

DETAILED DESCRIPTION:
Carfilzomib, lenalidomide and dexamethasone (CRD) combination therapy is generally associated with high response rates. The expectation is that induction therapy with CRD will result in responses within the myeloma lesions. Extrapolating from the published experience on standard bone marrow response rates with CRD regimen, it is predicted that guided biopsy of myeloma lesions will reveal VGPR/CR/nearCR rate up to 50%. Further, it can be hypothesized that myeloma lesion biopsy will increase the detection rate of residual/refractory disease by about 20%, as compared with standard bone marrow evaluation. Thus, it is expected that myeloma lesion biopsy response rate may be discordant from the standard bone marrow response rate. The identification of patients with large residual disease burden in the myeloma lesions will indicate the need for further salvage therapy. Based on this, it is expected that advanced imaging with guided myeloma lesion biopsy will result in significantly improved response assessment strategy after induction therapy, and will allow better selection of patients prior to autologous stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be diagnosed with symptomatic multiple myeloma within 90 days prior to registration
* Patients must have measurable or evaluable disease as defined by having one or more of the following, obtained within 35 days prior to randomization:
* Detectable monoclonal protein (M-protein) on serum protein electrophoresis
* Detectable monoclonal protein on a 24 hour urine protein electrophoresis
* Abnormal serum kappa to lambda free light chain ratio (< 0.26 or > 1.65)
* Clonal bone marrow plasma cells ≥10%
* Myeloma-defining bone lesion or extramedullary plasmacytoma on advanced imaging
* The following laboratory values must be obtained within 35 days prior to registration:
* Hemoglobin ≥ 7 g/dL
* Platelet count ≥ 50,000 cells/mm3
* Absolute neutrophil count ≥ 500 cells/mm3
* Calculated creatinine clearance ≥ 15 mL/min
* Bilirubin ≤ 2 mg/dL
* SGPT (ALT) and SGOT (AST) < 3 times the upper limit of normal. (Red blood cell and platelets transfusion is allowed to maintain the above goal) Patients may have received one cycle (28 days or less) of prior chemotherapy and no more than 320mg of prior dexamethasone (or equivalent dose of prednisone) for treatment of symptomatic myeloma. They may have received lenalidomide, bortezomib, or cyclophosphamide for treatment of symptomatic myeloma. They may not have received prior carfilzomib.
* Prior radiation therapy to symptomatic lesions is allowed provided 10 days is allowed between the completion of radiation therapy and start of protocol treatment.
* Prior systemic glucocorticoid use for the treatment of non-malignant disorders is permitted. Prior or concurrent topical or localized glucocorticoid therapy to treat non-malignant comorbid disorders is permitted.
* Patients must not have active, uncontrolled seizure disorder. Patients must have had no seizures in the last 6 months.
* Patients must not have uncontrolled concurrent illness including uncontrolled hypertension, symptomatic congestive heart failure, unstable angina, uncontrolled cardiac arrhythmia, uncontrolled psychiatric illness or social situation that would limit compliance with the study.
* ECOG performance status 0, 1, or 2. (PS 3 allowed if secondary to pain)
* Patients with monoclonal gammopathy of undetermined significance or asymptomatic multiple myeloma are not eligible.
* Patients must not have Grade 3 or higher peripheral neuropathy by CTCAE 4.0.
* Patients must not have active, uncontrolled infection requiring intravenous antibiotic therapy.
* Patients may have a history of current or previous deep vein thrombosis or pulmonary embolism but must be willing to receive anti-coagulation as prophylaxis if they are not currently on full-dose anticoagulation.
* Patients must not have New York Heart Association classification III or IV heart failure or myocardial infarction within the previous 6 months and must have left ventricular ejection fraction of at least 40%.
* Patients with a history of prior malignancy are eligible provided they were treated with curative intent and do not require active therapy (currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast are not excluded).
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 14 days prior starting lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, 14 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
* The patient must be able to undergo advanced imaging with either WB-MRI or PET scan.
* The patient must not have any inherited or acquired bleeding diathesis increasing the risk of hemorrhage with guided biopsies.
* HIV infection is not excluded. Known HIV positive patients must have documented CD4 cell count ≥ 350/mm3 and no history of AIDS-related illness.

Exclusion Criteria:

* Violation of inclusion criteria specifics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
Detection rate of residual/refractory | 4 months
  The purpose of this outcome is to compare standard biopsy procedures with the image guided approach. International Myeloma Working Group (IMWG) Criteria for Response and Progression standards will be used to determine the detection rate of residual/refractory.

SECONDARY OUTCOMES:
Myeloma lesion response rate | 4 months
  International Myeloma Working Group (IMWG) Criteria for Response and Progression standards will be used.
Overall clinical response rate | 4 months
  International Myeloma Working Group (IMWG) Criteria for Response and Progression standards will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Neparidze, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States